CLINICAL TRIAL: NCT07276737
Title: Preconditioning With a Combination of Thiotepa, Cyclophosphamide, and Busulfan for Allogeneic Hematopoietic Stem Cell Transplantation in the Treatment of NK/T-Cell Lymphoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Xianmin Song, MD, Director, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHSYXY-NT/T-TCB-2025
Record Dates: First submitted 2025-11-29; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: NK T-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell | interventions — Thiotepa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment group (Experimental)
  Interventions: Drug: Thiotepa

INTERVENTIONS:
Drug: Thiotepa — The enrolled patients began the pre-treatment on day d-9. The pre-treatment regimen was as follows: Thiotepa 5mg/kg/d, from -9d to -8d (2d); Cyclophosphamide: 40 - 50mg/kg/d, from -7d to -6d (2d); Busulfan injection: for patients under 55 years old with HCT-CI score of 2 or below, use 3.2mg/kg/d from -5d to -3d (3d), for those over 55 years old with HCT-CI score above 2, use 3.2mg/kg/d from -5d to -4d (2d);

SUMMARY:
Evaluation of the efficacy and safety of Thiotepa combined with Cyclophosphamide and Busulfan as conditioning regimen before allo-HSCT for the treatment of NK/T cell lymphoma

DETAILED DESCRIPTION:
Although allo-HSCT brings certain survival benefits to patients with NK/T cell lymphoma, post-transplantation relapse remains the main cause of treatment failure and death. Therefore, it is crucial to further optimize the pre-transplantation conditioning regimen. Thiotepa is a non-specific cell cycle drug with good anti-tumor effects; it also has the dual functions of myeloablative and immunosuppressive effects, which can increase the implantation success rate, reduce the incidence of GVHD and recurrence rate. Currently, Thiotepa has become one of the preferred drugs for pre-transplantation conditioning in patients with primary central nervous system lymphoma and acute lymphoblastic leukemia. This study aims to add Thiotepa to the commonly used RIC conditioning regimen in order to explore an efficient and low-toxicity pre-transplantation conditioning regimen for allo-HSCT in NK/T cell lymphoma patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age range: 18-70 years old, gender not restricted. 2. Patients diagnosed with NK/T cell lymphoma through histopathology or flow cytometry, 1) with stage III/IV patients receiving first-line or salvage treatment and achieving remission, 2) stage II patients with relapsed/refractory disease after salvage treatment achieving remission, 3) patients with NK cell lymphoma/leukemia receiving first-line or salvage treatment and achieving remission, 4) patients with relapsed/refractory disease. 3. Patients must have a suitable hematopoietic stem cell donor. 1) The related donor must have at least 5/10 HLA-A, -B, -C, -DQB1, and -DRB1 matching. 2) The unrelated donor must have at least 8/10 HLA-A, -B, -C, -DQB1, and -DRB1 matching. 4. HCT-specific comorbidity index score (HCT-CI) <= 2. 5. ECOG: 0-2 points. 6. Liver and kidney functions, as well as heart and lung functions, must meet the following requirements: 1) Serum creatinine <= 1.5 × ULN; 2) Cardiac function: Ejection fraction >= 50%; 3) Basal oxygen saturation > 92%; 4) Total bilirubin <= 1.5 × ULN; ALT and AST <= 2.0 × ULN; 5) Pulmonary function: DLCO (hemoglobin corrected) >= 40% and FEV1 >= 50%. 7. Patients must be capable of understanding and willing to participate in this study, and sign the informed consent form.

Exclusion Criteria:

1. Patients allergic to stietap, cyclophosphamide or busulfan or its components. 2. Any unstable systemic diseases: including but not limited to unstable angina pectoris, cerebrovascular accident or transient cerebral ischemia (within 3 months before screening), myocardial infarction (within 3 months before screening), congestive heart failure (NYHA classification ≥ III), severe arrhythmia requiring drug treatment, liver, kidney or metabolic diseases;patients with pulmonary hypertension. 3. Active and uncontrolled infections: hemodynamic instability related to infection, or new symptoms or signs of infection worsening, or new infection lesions found on imaging, persistent fever without exclusion of infection without symptoms or signs; 4. Grade 2 or higher epilepsy, paralysis, aphasia, new cerebral infarction, severe brain trauma, dementia, Parkinson's disease, schizophrenia 5. HIV-infected patients; 6. Patients with active hepatitis B (HBV) or active hepatitis C (HCV) requiring antiviral treatment; 2.patients with a risk of HBV activation, referring to those with positive hepatitis B surface antigen or core antibody but not receiving anti-hepatitis virus treatment; 7. Pregnant or lactating women; 8. Male and female individuals with reproductive capacity who are unwilling to use contraceptive methods during treatment and within 12 months after treatment; 9. Patients whose study investigators assess have other inadvisable inclusion conditions.

-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2029-12-30 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
progression free survival | Two years after the transplantation

SECONDARY OUTCOMES:
Cumulative recurrence rate | One year and two years after transplantation
Incidence of acute GVHD | within 180 days post-transplantation

IPD SHARING:
Plan to Share IPD: No